CLINICAL TRIAL: NCT07312643
Title: A Phase 1, Open-label, Randomized, Crossover Study in Healthy Subjects to Investigate the Relative Bioavailability and Safety of Pasireotide After Single Subcutaneous Dose Administration Using a Reusable ServoPen With Cartridge as Compared to Administration Using a Syringe Drawn From an Ampule
Brief Title: Study in Healthy Subjects to Investigate the Relative Bioavailability and Safety of Pasireotide After Single Subcutaneous Dose Administration Using a Reusable ServoPen With Cartridge as Compared to Administration Using a Syringe Drawn From an Ampule
Acronym: PASIPHY_PEN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Collaborators: Nuvisan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SOM230-RECAG-PK-0605
Record Dates: First submitted 2025-11-19; First posted 2025-12-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pharmacokinetics; Safety
Keywords: pasireotide; subcutaneous; bioavailability
MeSH Terms: interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ServoPen 50 µg (Experimental): Single dose of 50 µg pasireotide administered subcutaneously using reusable ServoPen with cartridge.
  Interventions: Combination Product: Pasireotide cartridge with reusable ServoPen
- ServoPen 200 µg (Experimental): Single dose of 200 µg pasireotide administered subcutaneously using reusable ServoPen with cartridge.
  Interventions: Combination Product: Pasireotide cartridge with reusable ServoPen
- Syringe 50 µg (Active Comparator): Single dose of 50 µg pasireotide administered subcutaneously using syringe drawn from an ampule.
  Interventions: Drug: Pasireotide ampule with syringe
- Syringe 200 µg (Active Comparator): Single dose of 200 µg pasireotide administered subcutaneously using syringe drawn from an ampule.
  Interventions: Drug: Pasireotide ampule with syringe

INTERVENTIONS:
Combination Product: Pasireotide cartridge with reusable ServoPen — Pasireotide cartridge with reusable ServoPen
  Arms: ServoPen 200 µg; ServoPen 50 µg
Drug: Pasireotide ampule with syringe — Pasireotide ampule with syringe
  Arms: Syringe 200 µg; Syringe 50 µg

SUMMARY:
This single-center Phase 1 study in healthy male and female subjects of 18 to 55 years (inclusive) will follow an open-label, randomized, single-dose, crossover design with 2 intervention periods. The purpose of this study is to assess and compare the pharmacokinetic characteristics and the safety of single doses of pasireotide when administered subcutaneously by reusable ServoPen with cartridge or by syringe drawn from an ampule in healthy subjects.

DETAILED DESCRIPTION:
Study details include:

* The study duration will be approximately 6.5 weeks per subject.
* Two (2) intervention periods are planned per dose level (50 µg and 200 µg), with 1 of the following interventions administered per period:

  * Single dose of 50 µg pasireotide administered subcutaneously using reusable ServoPen with cartridge.
  * Single dose of 200 µg pasireotide administered subcutaneously using reusable ServoPen with cartridge.
  * Single dose of 50 µg pasireotide administered subcutaneously using syringe drawn from an ampule.
  * Single dose of 200 µg pasireotide administered subcutaneously using syringe drawn from an ampule.
* The screening examination will be performed within 28 to 2 days prior to the first administration of study intervention.
* Subjects will stay in-house for at least 3 days per period.
* The ambulatory follow-up visit will be performed within 7 to 10 days after the last administration of study intervention.

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible only if all of the following criteria apply:

  1. Age of 18 to 55 years inclusive, at the time of signing the informed consent.
  2. BMI ≥18.5 kg/m2.
  3. Male or female. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

     a. Male subjects: Male subjects are eligible to participate if they agree to the following starting from the first administration of study intervention until the follow-up visit:

     • Refrain from donating semen. Plus, either:

     o Abstain from sexual intercourse with a partner of childbearing potential (definition in Section 10.5.1 of Study Protocol (SP)). OR

     o During sexual intercourse with a partner of childbearing potential, use a male condom and counsel the partner to use a highly effective contraceptive method (definitions in Section 10.5.2 of SP).

     b. Female subjects: A female subject is eligible to participate if she is neither pregnant nor breastfeeding, and one of the following conditions applies:

     • Postmenopausal or has been sterilized more than 3 months ago (definitions in Section 10.5.1 of SP). OR

     • Uses a highly effective (with a failure rate of <1% per year) contraceptive method, preferably with low user dependency, as described in Section 10.5.2 during study participation and for at least 30 days after the last administration of study intervention and agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.

     ❑General Health Status
  4. Overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs and ECG.
  5. Clinically acceptable clinical laboratory test results.

     ❑Smoking
  6. Non-smoker, which includes abstinence from using other nicotine-containing products (e.g., nicotine patches, chewing gum, e-cigarettes) for at least the last 3 months prior to first administration of study intervention.

     * Informed Consent
  7. Capable of giving signed informed consent as described in Section 10.1 of SP, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol prior to any clinical study-specific procedure.

     EXLCUSION:

     Subjects are excluded from the study if any of the following criteria apply:
     * Medical Conditions

  <!-- -->

  1. Any history or evidence of any clinically relevant and/or other major disease or malignancy as determined by medical evaluation (including physical examination) capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention or interfering with the interpretation of data.
  2. Contraindications for the use of pasireotide in medical history, such as ≥ moderate hepatic impairment (Child-Pugh B), hypocortisolism, uncontrolled diabetes, heart failure ≥ New York Heart Association Class III, cardiogenic shock, second- or third-degree AV block, sinoatrial block, sick sinus syndrome, severe bradycardia or congenital long QT syndrome.
  3. Medical history of pituitary disorder.
  4. History or presence of cholelithiasis and/or acute or chronic pancreatitis.
  5. Any clinically relevant history of allergic conditions requiring hospitalization or prolonged systemic treatment (including drug allergies, drug hypersensitivity, asthma, eczema, allergies requiring therapy with corticosteroids or anaphylactic reactions), excluding allergic contact sensitizations (e.g., nickel allergy). Subjects with uncomplicated seasonal allergic rhinitis can be accepted if the expected allergy season is clearly outside the study period.
  6. Known or suspected hypersensitivity to study interventions or any component of the formulations used.
  7. Clinically relevant chronic or acute infectious illness or febrile illness within the last 14 days prior to first administration of study intervention.
  8. Evidence of COVID-19 signs or symptoms or confirmed COVID-19 infection within the last 14 days prior to first administration of study intervention.
  9. Tendency for vasovagal reactions (e.g., after venipuncture) or history of syncope.

     * Diagnostic Assessments
  10. Positive for hepatitis B surface antigen, hepatitis C antibody or anti-HIV 1 + 2 antibodies and HIV 1 p24 antigen.
  11. Positive test for alcohol or drugs of abuse.
  12. Positive pregnancy test in female subjects.
  13. Supine systolic blood pressure >140 mmHg or 90 mmHg or 90 bpm or tympanic body temperature 37.6°C.
  14. 12-lead ECG with clinically relevant abnormality or showing a QTcF>450 ms for male or >470 ms for female subjects, PR >215 ms or QRS >120 ms.
  15. Fasting glucose ≥ 5.5 mmol/L at screening and/or HbA1c > ULN at screening.
  16. ALT ≥1.5 x ULN, AST ≥1.5 x ULN or serum bilirubin ≥1.5 x ULN.
  17. eGFR calculated based on the Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation
  18. Thyroid disorders as evidenced by TSH outside normal range and confirmed by free triiodothyronine and free thyroxine outside normal range. Subjects with suspected compensated thyroid hormone formation disorders as indicated by TSH outside normal range but free triiodothyronine and free thyroxine within normal range may be included at the discretion of the Investigator.
  19. Hypokalemia (potassium ≤ 3.5 mmol/L).
  20. Hypomagnesemia (magnesium < 0.7 mmol/L).

      ❑Prior/Concomitant Therapy
  21. Use of any concomitant medication or any drugs / medicines (including dietary supplements, natural and herbal remedies) within the last 14 days or 5 times their elimination half-life prior to first administration of study intervention, whichever is longer. Allowed treatments are the use of contraceptives as outlined in Section 10.5 of SP and HRT if the subject has been on stable treatment for at least 3 months and continues treatment throughout the study. Additionally, the occasional use of paracetamol (up to 2 g per day) and ibuprofen (up to 1.6 g per day) are allowed.

      ❑Prior/Concurrent Clinical Study Experience
  22. Use of any investigational drug or participation in any clinical study within 30 days or 5 times the half-life of the study drug administered in a previous study, whichever is longer, prior to the expected date of first administration of study intervention.
  23. Previous randomization in this study.

      ❑Other Exclusions
  24. Higher than low-risk alcohol consumption i.e., consumption of an average weekly alcohol intake of >14 units/week for men (daily dose of >24 g, weekly dose of >168 g) and >7 units/week for women (daily dose of >12 g, weekly dose of >84 g). One unit (12 g) corresponds to 0.3 L of beer/day or 0.12 L of wine/day or 2 cL of spirits/day.
  25. History of drug or alcohol abuse within the last 6 months.
  26. Excessive consumption of caffeine- or xanthine-containing food or beverages (>5 cups of coffee a day or equivalent) or inability to stop consuming within 48 h prior to planned administration of study intervention
  27. Intake of food, beverages, or other products containing grapefruit, grapefruit juice, grapefruit hybrids, star fruit, Seville orange, tangelo, pomelo, or exotic citrus fruits within 14 days prior to planned administration of study intervention.
  28. Consumption of poppy seed containing food within the last 72 h prior to the first administration of study intervention.
  29. Vegetarian, vegan, or restricted diet (e.g., gluten-free) or not willing or able to eat the standard meals provided.
  30. Donation or blood collection of more than 450 mL of blood or blood products or acute loss of blood within the last 30 days prior to the first administration of study intervention.
  31. Strenuous physical activity within the last 72 h prior to the first administration of study intervention.
  32. Employee of the Sponsor, the Nuvisan Group, or other CRO involved in the clinical study.
  33. Legal incapacity or limited legal capacity, or incarceration.
  34. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the protocol requirements, instructions, and study-related restrictions.
  35. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-03 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
AUC0-tlast | 2 weeks
  To investigate the relative bioavailability (Frel) of pasireotide s.c. after single-dose administration of 2 dose levels using reusable ServoPen with cartridge (Test 1 and Test 2) compared to single-dose administration of 2 dose levels using syringe drawn from an ampule (Reference 1 and Reference 2).
AUC0-inf | 2 weeks
  To investigate the relative bioavailability (Frel) of pasireotide s.c. after single-dose administration of 2 dose levels using reusable ServoPen with cartridge (Test 1 and Test 2) compared to single-dose administration of 2 dose levels using syringe drawn from an ampule (Reference 1 and Reference 2).
Cmax | 2 weeks
  To investigate the relative bioavailability (Frel) of pasireotide s.c. after single-dose administration of 2 dose levels using reusable ServoPen with cartridge (Test 1 and Test 2) compared to single-dose administration of 2 dose levels using syringe drawn from an ampule (Reference 1 and Reference 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan GmBH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No